CLINICAL TRIAL: NCT03081520
Title: Affective Responses Following Aerobic Exercise With Different Intensities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Affective responses exercise
Record Dates: First submitted 2017-03-07; First posted 2017-03-16 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2017-07

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Affective response MIT (Experimental): Moderate intensity continuous training 50 min with walking or running on approximately 75% of HRmax
  Interventions: Behavioral: Affective response MIT
- Affective response HAIT (Experimental): High-Intensity Aerobic Interval Training 4x4 min with walking or running on 85-95% of HRmax 3 min active recovery between sets, intensity of approximately 70% of HRmax
  Interventions: Behavioral: Affective response HAIT
- Affective response HIIT (Experimental): High-Intensity Interval Training 4-6 x 30-sec sprints on tread mill, >95% HRmax during sprints 4 min recovery between sprints, intensity of approximately 70% of HRmax
  Interventions: Behavioral: Affective response HIIT

INTERVENTIONS:
Behavioral: Affective response MIT — Examine acute affective responses during and after five sessions of endurance training with moderate intensity continuous training
  Arms: Affective response MIT
Behavioral: Affective response HAIT — Examine acute affective responses during and after five sessions of endurance training with high-intensity aerobic interval training
  Arms: Affective response HAIT
Behavioral: Affective response HIIT — Examine acute affective responses during and after five sessions of endurance training with high-intensity sprint interval training
  Arms: Affective response HIIT

SUMMARY:
The aim of this study is to examine acute affective responses during and after a series of exercise sessions with different intensities in young healthy adults. The study is a randomized controlled trial with three different groups (A: moderate continuous training (MIT), B: high-intensity aerobe interval training (HAIT), C: high-intensity sprint interval training (HIIT)). Healthy adults aged 18-40 years (n=30) will be invited to participate. Each participant will perform a VO2max test followed by five session of the randomized type of training. The sessions will be completed within two weeks. The participants will complete questionnaires regarding exercise motivation (Behavioral Regulation of Exercise Questionnaire), mood (Positive and Negative Affect Scale, Profile of Mood States, Visual Analogue scale, Self-assessment Manikin Rating Scale) and perceived exhaustion (Borg Ratings of Perceived Exertion scale). In addition, blood lactate and heart rate will be obtained during and after each session.

DETAILED DESCRIPTION:
Physical activity has is considered as one of the most important health related aspects of the 21st century. In Norway, large epidemiological studies show that only about 30% of the adult population meet the physical activity recommendations of 150 minutes per week with moderate-to-vigorous intensity physical activity. Also, studies show that there are large dropout rates from lifestyle interventions, and that approximately 50% drop out from physical activity interventions within 6 months after start. One explanation for the dropout is performance of exercise with too vigorous intensities.

Very vigorous intensity physical activity can be experienced as unpleasant. According to the dual-mode theory there are positive affective responses after low-to-moderate intensity physical activity, whereas vigorous intensity physical activity trigger negative affective responses which again can lead to reduced motivation for the exercise. Unfortunately, many of the studies performed on affective responses to exercise have used one session only. The studies who have examined changes in affective responses after series of exercise have used vigorous intensities above the anaerobic threshold, and it is therefore unknown whether similar affective responses occur in vigorous intensity aerobe exercise.

The aim of this study is to examine acute affective responses during and after a series of exercise sessions with different intensities in young healthy adults.

To examine this, a randomized controlled clinical trial with three different groups (moderate intensity training (MIT), high-intensity aerobic interval training (HAIT) and high-intensity sprint interval training (HIIT)) will be conducted. A power calculation showed need for recruitment of 30 participants. The sample will consist of healthy young adults. All participants will perform one VO2max test, and five sessions with the intensity they are randomized to. All six sessions (test + exercise sessions) will be conducted within two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No high intensity interval training during the past three months prior to participation
* Regular exercise up to two sessions per week
* 18-40 years of age
* BMI <30 kg/m2

Exclusion Criteria:

* Competing athlete
* Smoker
* Injury not compatible with performing the exercises
* BMI <16 kg/m2
* Pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change in self rated well-being rated on a Visual Analogue Scale | Two weeks
  well-being rated on a Visual Analogue Scale

SECONDARY OUTCOMES:
Self-reported change in affects using Positive and Negative Affect Scale | Two weeks
  Positive and Negative Affect Scale
Self-reported change in physical activity motivation using Behavioural Regulation of Exercise Questionnaire - 2 | Two weeks
  Behavioural Regulation of Exercise Questionnaire - 2
Self-reported change in affective responses using Self-Assessment Manikin Rating Scale | Two weeks
  Self-Assessment Manikin Rating Scale
Self-reported change in mood using scale Profile of Mood States | Two weeks
  Use of the standardized and validated scale Profile of Mood States
Perceived exercise intensity during each exercise session using Borgs Ratings of Perceived Exertion (RPE) scale (6-20) | At minutes 0,10, 20, 40 and 50 in each exercise session
  Borgs RPE scale (6-20)
Lactate during each exercise session (mMol/l) | At minutes 0,10, 20, 40 and 50 in each exercise session
  Blood lactate samples (mMol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Solfrid Bratland-Sanda, PhD, Principal Investigator — University College of Southeast Norway
Locations (1):
- University College of Southeast Norway, Bø, Telemark, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saanijoki T, Nummenmaa L, Eskelinen JJ, Savolainen AM, Vahlberg T, Kalliokoski KK, Hannukainen JC. Affective Responses to Repeated Sessions of High-Intensity Interval Training. Med Sci Sports Exerc. 2015 Dec;47(12):2604-11. doi: 10.1249/MSS.0000000000000721. PMID 26110694
- [Background] Ekkekakis P, Parfitt G, Petruzzello SJ. The pleasure and displeasure people feel when they exercise at different intensities: decennial update and progress towards a tripartite rationale for exercise intensity prescription. Sports Med. 2011 Aug 1;41(8):641-71. doi: 10.2165/11590680-000000000-00000. PMID 21780850
- [Background] Williams DM. Exercise, affect, and adherence: an integrated model and a case for self-paced exercise. J Sport Exerc Psychol. 2008 Oct;30(5):471-96. doi: 10.1123/jsep.30.5.471. PMID 18971508